CLINICAL TRIAL: NCT02478736
Title: Preoperative Transcranial Doppler as a Predictor for Delirium Following On-pump Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0319
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Delirium After On-pump Cardiac Surgery
Keywords: postoperative delirium; on-pump cardiac surgery; cerebral oximetry; cerebral blood flow velosity
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- delirium group: the patients with delirum after on-pump cardiac surgery
  Interventions: Other: No actual intervention
- no delirium group: the patients without delirum after on-pump cardiac surgery
  Interventions: Other: No actual intervention

INTERVENTIONS:
Other: No actual intervention — Contact with enrolled subjects requires application of ceberal oximetry electrodes and the preoperative ultrasound (transcranial doppler) of the both MCA. No actual intervention done to subject.

SUMMARY:
Postoperative delirium is an important problem in patients undergoing major cardiac surgery and associated with more complicated hospital course, increased hospital length of stay and total postoperative cost. A study shows that a low preoperative cerebral oximetry (rSO2) is associated with postoperative delirium after on-pump cardiac surgery. Another study showed that patients who underwent cardiac surgery with reduced cerebral blood flow (CBF) velocity in the left middle cerebral artery (MCA) preoperatively are at greater risk for postoperative cognitive dysfunction (POCD). Therefore, the investigators hypothesize that lower perioperative rSO2 and reduced preoperative mean flow velocity (MFV) of MCA are good predictors of the postoperative delirium in the patients undergoing the on-pump cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the study will be 60 or older undergoing elective major on-pump cardiac surgery

Exclusion Criteria:

1. No communication possible due to a language barrier or deafness
2. Patients diagnosed with neurocognitive disorders or psychiatric diseases (MMSE or Geriatric Depression Scale cannot be checked before surgery)
3. Patients with unstable hemodynamics or intubated before surgery
4. Patients diagnosed with significant (≥ 50%) intracranial stenosis confirmed by CT angiography or MR angiography
5. Patients diagnosed with stroke, TIA or neurologic diseases (e.g. Parkinson's disease, epilepsy, dementia, or taking psychiatric medications d/t psychiatric disorders)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing on-pump cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
the predictive power of perioperative MFV of MCA regarding postoperative delirium | 7 days from postoperation
  The presence and severity of delirium were assessed with Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) once a day. The investigators plan to evaluate whether perioperative rSO2 and/or MFV of MCA can predict postoperative delirium in patients undergoing the on-pump cardiac surgery and to assess the predictive power of perioperative rSO2/MFV of MCA regarding postoperative delirium. Perioperative rSO2 was observed during surgery (an expected average of 4 hours) and MVF of MCA was measured just before the induction of general anesthesia.
the predictive power of periopertiver rSO2 values regarding postoperative delirium | 7 days from postoperation
  To evaluate whether periopertiver MFV of MCA and/or rSO2 can predict postoperative delirium in patients undergoing the on-pump cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea